CLINICAL TRIAL: NCT00004072
Title: Phase II Trial of O6-Benzylguanine (NSC 637037) and BCNU in Patients With Multiple Myeloma
Brief Title: O6-benzylguanine And Carmustine in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Stanton L. Gerson, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1A96; U01CA062502 (NIH); P30CA043703 (NIH); CWRU-1A96 (Other: Case Comprehensive Cancer Center); NCI-T97-0021
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — O(6)-benzylguanine; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: O6-benzylguanine — Patients receive O6-benzylguanine IV over 60 minutes. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients receive 2 additional courses beyond attainment of best response.
Drug: carmustine — Followed 1 hour later by carmustine IV over 60 minutes. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients receive 2 additional courses beyond attainment of best response.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining O6-benzylguanine with carmustine in treating patients who have previously untreated, refractory, or relapsing multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy of O6-benzylguanine combined with carmustine in patients with previously untreated or refractory multiple myeloma.
* Assess the effects of O6-benzylguanine on bone marrow myeloma cells in this patient population.

OUTLINE: Patients receive O6-benzylguanine IV over 60 minutes followed 1 hour later by carmustine IV over 60 minutes. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients receive 2 additional courses beyond attainment of best response (partial or complete response or stable or plateau disease).

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed progressive multiple myeloma, meeting 1 of the following criteria:

  * Previously untreated
  * Primary refractory
  * Relapsing disease
* Major criteria:

  * Plasmacytomas on tissue biopsy
  * Bone marrow plasmacytosis with greater than 30% plasma cells
  * Monoclonal globulin spike on serum electrophoresis

    * Greater than 3.5 g/dL for G peaks or greater than 2.0 g for A peaks
    * Greater than 1.0 g/24 hours of kappa or lambda light chain excretion on urine electrophoresis in the absence of amyloidosis
* Minor criteria:

  * 10%-30% bone marrow plasmacytosis (criterion A)
  * Presence of monoclonal globulin spike but less than the levels under major criteria (criterion B)
  * Lytic bone lesions (criterion C)
  * IgM less than 50 mg/dL, IgA less than 100 mg/dL, or IgG less than 600 mg/dL (criterion D)
* Must meet one of the following:

  * A minimum of 1 major criterion and 1 minor criterion
  * 3 minor criteria, including criteria A and B

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3
* Absolute neutrophil count greater than 1,500/mm^3
* Hemoglobin greater than 9 g/dL (transfusions allowed)

Hepatic:

* Bilirubin less than 1.5 mg/dL
* AST/ALT less than 2 times normal

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance greater than 60 mL/min
* Calcium less than 14 mg/dL

Pulmonary:

* No prior or concurrent active, symptomatic respiratory disease
* Corrected DLCO at least 60% predicted

Other:

* Controlled diabetes mellitus allowed
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No more than 1 prior chemotherapy regimen containing an alkylating agent for multiple myeloma
* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Prior corticosteroids for multiple myeloma allowed

Radiotherapy:

* No prior pelvic radiotherapy or radiotherapy to more than 25% of bone marrow

Surgery:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 1999-09; Primary Completion 2004-08 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of O6-benzylguanine combined with carmustine in patients with previously untreated or refractory multiple myeloma. | Every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients receive 2 additional courses beyond attainment of best response. Patients are followed every 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: Stanton L. Gerson, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio